CLINICAL TRIAL: NCT03886519
Title: Repeat Surgery for Patients With Post-operative Trachomatous Trichiasis Trial
Acronym: PTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Orbis (Other); National Eye Institute (NEI) (NIH); University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-2766; UG1EY025992-04S1 (NIH)
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Results first posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2022-08

CONDITIONS: Trichiasis; Surgery
MeSH Terms: conditions — Trichiasis | interventions — Inosine Monophosphate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRAP (Bevel/rotate/advance procedure) (Active Comparator): The BRAP procedure is a full-thickness beveled full-thickness incision
  Interventions: Procedure: BRAP (Bevel/rotate/advance procedure)
- Trabut 3 mm (Active Comparator): The Trabut procedure is a partial-thickness incision through the tarsal conjunctiva and tarsus parallel to the eyelid margin and 3 mm above the lash line.
  Interventions: Procedure: Trabut

INTERVENTIONS:
Procedure: BRAP (Bevel/rotate/advance procedure) — Trichiasis surgery using the BRAP procedure
  Other Names: BRAP procedure
  Arms: BRAP (Bevel/rotate/advance procedure)
Procedure: Trabut — Trichiasis surgery using the Trabut procedure
  Other Names: Trabut procedure
  Arms: Trabut 3 mm

SUMMARY:
The objective of this study is to determine if there is a significant difference in post-operative trichiasis at 12 months comparing a new procedure, the Bevel/rotate/advance procedure (BRAP), to the Trabut procedure among repeat surgery patients.

DETAILED DESCRIPTION:
The investigators will randomize participants with previously operated trichiasis on a 1:1 basis to receive either the Bevel/rotate/advance procedure (BRAP) or the Trabut procedure. The participants will be followed at 1 day, 2 weeks, 3-6 months, and then 12 months following the surgery. The primary study endpoint is recurrence of post-operative trichiasis within 12 months of surgery. The investigators will conduct logistic regression analysis comparing post-operative trichiasis recurrent rates in participants receiving BRAP versus participants receiving Trabut. Adjusted analyses will account for demographic characteristics as well as trichiasis severity prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* At least one eyelid with post-operative upper eyelid trichiasis
* Willing to comply with all study procedures and be available for the duration of the study

Exclusion Criteria:

* Inability to provide independent, informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 886 (Actual)
Dates: Start 2019-04-13 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2022-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Gower, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Orbis Ethiopia, Hosa’ina, Southerns Nations, Nationalities, and Peoples' Region, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made available at the time of publication of the primary and pre-planned secondary results papers.
Supporting Information: Study Protocol, SAP
Time Frame: Deidentified individual data that support the results will be shared beginning 9 to 36 months following publication.
Access Criteria: An investigator who proposes to use the data must have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and execute a data use/sharing agreement with UNC.

REFERENCES:
- [Background] Gower EW, West SK, Cassard SD, Munoz BE, Harding JC, Merbs SL. Definitions and standardization of a new grading scheme for eyelid contour abnormalities after trichiasis surgery. PLoS Negl Trop Dis. 2012;6(6):e1713. doi: 10.1371/journal.pntd.0001713. Epub 2012 Jun 26. PMID 22745845

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 886 participants were enrolled. Of those enrolled, 700 received surgery in accordance with the surgical protocol and the analyses are based on these participants.
Units Other Than Participants: Eyes
Groups:
- BRAP (Bevel/Rotate/Advance Procedure): The Bevel/rotate/advance procedure (BRAP) involves a partial-thickness beveled incision and tarsal advancement.
  BRAP: Trichiasis surgery using the BRAP procedure
Period: Overall Study
Arm/Group | BRAP (Bevel/Rotate/Advance Procedure) | Trabut 3 mm
Started | 351; 446 Eyes | 349; 446 Eyes
3-6 Month Visit | 264; 317 Eyes | 252; 337 Eyes
12 Month Visit | 312; 399 Eyes | 316; 399 Eyes
Completed (Primary outcomes based on completing either the 3-6 month visit and/or the 12 month visit. Therefore, number completed is greater than the number of individuals seen at either visit.) | 335; 425 Eyes | 328; 420 Eyes
Not Completed | 16; 21 Eyes | 21; 26 Eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- BRAP (Bevel/Rotate/Advance Procedure): The BRAP procedure involves a partial-thickness beveled incision, tarsal advancement and rotation
  BRAP (Bevel/rotate/advance procedure): Trichiasis surgery using the BRAP procedure
- Total: Total of all reporting groups
Arm/Group | BRAP (Bevel/Rotate/Advance Procedure) | Trabut 3 mm | Total
Number analyzed (Participants) | 351 | 349 | 700
Number analyzed (Eyes) | 446 | 446 | 892
Age, Customized [Count of Participants; unit: Participants]
  <40 years | 92 | 75 | 167
  40-60 years | 189 | 193 | 382
  >60 years | 70 | 81 | 151
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 285 | 273 | 558
  Male | 66 | 76 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 351 | 349 | 700
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 351 | 349 | 700
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Ethiopia | 351 | 349 | 700
Baseline Trachomatous Trichiasis (TT) Severity [Count of Units; unit: Eyes] — Trichiasis severity will be graded as mild, moderate, or severe based on number of eyelashes touching globe and number of eyelashes epilated. Definitions: Mild: 1-4 Eyelashes touching globe, no epilation OR 1-10 Eyelashes epilated, no eyelashes touching globe; Moderate: 5-9 Eyelashes touching globe, no epilation OR 1-4 Eyelashes touching globe and 1-10 eyelashes epilated; Severe: 5-9 Eyelashes touching globe and 1-10 eyelashes epilated OR 10+ Eyelashes touching globe, regardless of epilation status OR 11-20 Eyelashes epilated, regardless of eyelashes touching globe OR Entire eyelid epilated
  Eyes
    Mild | 74 | 74 | 148
    Moderate | 84 | 104 | 188
    Severe | 288 | 268 | 556

OUTCOME MEASURES:

1. Primary Outcome: Number of Eyelids With Post-operative Trichiasis Within 12 Months
Description: Presence of post-operative trichiasis defined as at least one trichiatic eyelashes or evidence of recent epilation. Trichiatic eyelashes are eyelashes touching the globe with the eye in the primary gaze. The outcome will be assessed at 3-6 months and at 12 months. If the eyelid has trichiasis at 2 weeks, but not at 3-6 months or 12 months, the eyelid will not be considered to have post-operative trichiasis. Due to COVID, the visit window for the Month 12 visits ranged from 10-20 months.
Time Frame: 10-20 months
Population: Data reported for those participants who completed the Month 3-6 and/or Month 12 assessments. A participant could have one or two eyes eligible for the study based on the number of eyes with TT prior to surgery.
Measure: Count of Units; unit: Eyelids
Units Other Than Participants: Eyelids
Groups:
- BRAP (Bevel/Rotate/Advance Procedure): The BRAP procedure is a partial-thickness beveled incision
  BRAP (Bevel/rotate/advance procedure): Trichiasis surgery using the BRAP procedure
Arm/Group | BRAP (Bevel/Rotate/Advance Procedure) | Trabut 3 mm
Number analyzed (Participants) | 335 | 328
Number analyzed (Eyelids) | 425 | 420
Eyelids | 94 | 120
Statistical Analysis 1: Comparison: BRAP (Bevel/Rotate/Advance Procedure) vs Trabut 3 mm; Test type: Superiority; p = 0.07, Regression, Logistic — The a priori threshold for statistical significance is <0.05; Adjusted for correlation between 2 eyes of a participant and baseline trichiasis severity; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.52 to 1.03]

2. Secondary Outcome: Number of Eyelids With Presence of Post-operative Trichiasis Within 3-6 Months
Description: Presence of post-operative trichiasis defined as at least one trichiatic eyelash or evidence of recent epilation. Trichiatic eyelashes are eyelashes touching the globe with the eye in primary gaze.
Time Frame: 3-6 months
Measure: Count of Units; unit: Eyelids
Units Other Than Participants: Eyelids
Arm/Group | BRAP (Bevel/Rotate/Advance Procedure) | Trabut 3 mm
Number analyzed (Participants) | 264 | 252
Number analyzed (Eyelids) | 317 | 337
Eyelids | 33 | 49

3. Secondary Outcome: Number of Eyelids With Each of the Trichiasis Severity Levels at 3-6 Months
Description: Severity will be graded as mild, moderate, or severe based on the number of eyelashes touching the globe and the amount of eyelashes epilated.
  Trichiasis severity will be defined using the following categories:
  i. Mild: 1-4 eyelashes touching globe and no epilation OR <1/3 eyelashes epilated and no eyelashes touching the globe ii. Moderate: 5-9 eyelashes touching globe and no epilation OR 1-4 eyelashes touching globe and <1/3 eyelashes epilated iii. Severe: 5-9 eyelashes touching globe and <1/3 eyelashes epilated OR 10+ eyelashes touching globe (regardless of epilation status) OR ≥1/3 eyelashes epilated (regardless of eyelashes touching globe) OR entire eyelid epilated
Time Frame: 3-6 months
Measure: Count of Units; unit: Eyelids
Units Other Than Participants: Eyelids
Arm/Group | BRAP (Bevel/Rotate/Advance Procedure) | Trabut 3 mm
Number analyzed (Participants) | 264 | 252
Number analyzed (Eyelids) | 317 | 337
Eyelids
  None | 284 | 288
  Mild | 21 | 32
  Moderate | 7 | 11
  Severe | 5 | 6

4. Secondary Outcome: Number of Eyelids With Each of the Trichiasis Severity Levels at 12 Months
Description: Severity will be graded as mild, moderate, or severe based on the number of eyelashes touching the globe and the amount of eyelashes epilated.
  Trichiasis severity will be defined using the following categories:
  i. Mild: 1-4 eyelashes touching globe and no epilation OR <1/3 eyelashes epilated and no eyelashes touching the globe ii. Moderate: 5-9 eyelashes touching globe and no epilation OR 1-4 eyelashes touching globe and <1/3 eyelashes epilated iii. Severe: 5-9 eyelashes touching globe and <1/3 eyelashes epilated OR 10+ eyelashes touching globe (regardless of epilation status) OR ≥1/3 eyelashes epilated (regardless of eyelashes touching globe) OR entire eyelid epilated.
  Due to COVID, the visit window for the Month 12 visits ranged from 10-20 months.
Time Frame: 10-20 months
Measure: Count of Units; unit: Eyelids
Units Other Than Participants: Eyelids
Arm/Group | BRAP (Bevel/Rotate/Advance Procedure) | Trabut 3 mm
Number analyzed (Participants) | 312 | 316
Number analyzed (Eyelids) | 399 | 399
Eyelids
  None | 310 | 281
  Mild | 47 | 76
  Moderate | 24 | 23
  Severe | 18 | 19

5. Secondary Outcome: Change in Severity of Post-operative Trichiasis Between 3-6 Months and 1 Year Using Grading System
Description: The change in PTT severity between 3-6 months and 12 months will be measured in eyes with PTT at 3-6 months that also were examined at the 12-month visit. Change will be measured in the difference in the number of categories between 3-6 month and 1 year outcome. For example, Mild to Severe would be a 2 category change.
Time Frame: 10-20 months
Population: Analysis limited to eyelids with PTT at 3-6 months that also had a 12-month visit.
Measure: Count of Units; unit: Eyelids
Units Other Than Participants: Eyelids
Arm/Group | BRAP (Bevel/Rotate/Advance Procedure) | Trabut 3 mm
Number analyzed (Participants) | 24 | 40
Number analyzed (Eyelids) | 28 | 47
Eyelids
  No change | 21 | 43
  1 category worse | 6 | 1
  2 categories worse | 1 | 3

6. Secondary Outcome: Number of Eyelids With Moderate/Severe Eyelid Contour Abnormalities at 3-6 Months
Description: The examiner will assess for eyelid contour abnormalities (ECA) and grade the abnormalities as mild, moderate, or severe. For the analysis, no abnormality and mild eyelid contour abnormality will be combined, and moderate and severe eyelid contour abnormality will be combined. For secondary analyses, the investigators will classify eyelid contour abnormalities using the photographs to capture the full range of ECA categories: none, mild, moderate, and severe.
  The definitions for the categories are: 1) Mild: Vertical deviation from the natural contour, 1 mm in height (less than half the pupil height in daylight) and affecting 1/3 of horizontal eyelid length. 2) Moderate: Vertical deviation from the natural contour 1-2 mm in height (about the pupil height in daylight) or affecting 1/3-2/3 of horizontal eyelid length 3) Severe: Vertical deviation from the natural contour 2 mm in height (more than the pupil height in daylight) or a defect >2/3 of the horizontal eyelid len
Time Frame: 3-6 months
Measure: Count of Units; unit: Eyelids
Units Other Than Participants: Eyelids
Arm/Group | BRAP (Bevel/Rotate/Advance Procedure) | Trabut 3 mm
Number analyzed (Participants) | 264 | 252
Number analyzed (Eyelids) | 317 | 337
Eyelids
  None/Mild | 225 | 236
  Moderate/Severe | 92 | 101

7. Secondary Outcome: Number of Eyelids With Moderate/Severe Eyelid Contour Abnormalities at 12 Months
Description: The examiner in the field will assess for eyelid contour abnormalities and grade the abnormalities as mild, moderate, or severe. For the analysis, no abnormality and mild eyelid contour abnormality will be combined, and moderate and severe eyelid contour abnormality will be combined. For secondary analyses, the investigators will classify eyelid contour abnormalities using the photographs to capture the full range of ECA categories: none, mild, moderate, and severe.
  The definitions for the categories are: 1) Mild: Vertical deviation from the natural contour, 1 mm in height (less than half the pupil height in daylight) and affecting 1/3 of horizontal eyelid length. 2) Moderate: Vertical deviation from the natural contour 1-2 mm in height (about the pupil height in daylight) or affecting 1/3-2/3 of horizontal eyelid length 3) Severe: Vertical deviation from the natural contour 2 mm in height (more than the pupil height in daylight) or a defect >2/3 of the horizontal eyelid length
Time Frame: 10-20 months
Measure: Count of Units; unit: Eyelids
Units Other Than Participants: Eyelids
Arm/Group | BRAP (Bevel/Rotate/Advance Procedure) | Trabut 3 mm
Number analyzed (Participants) | 312 | 316
Number analyzed (Eyelids) | 399 | 399
Eyelids
  None/Mild | 317 | 334
  Moderate/Severe | 82 | 65

8. Secondary Outcome: Cumulative Number of Eyelids With Presence of Pyogenic Granulomas Within 10-20 Months
Description: Pyogenic granulomas occasionally develop after trichiasis surgery. It is thought that this is a response to a foreign material, such as a sutures or an incision edge. All granulomas will be noted regardless of size. The investigators will count granulomas observed at the 3-6 month visit (including participants where the granuloma was removed) and granulomas observed at the 12 month visit. Due to COVID, the visit window for the Month 12 visits ranged from 10-20 months.
Time Frame: 10-20 months
Population: as for outcome 1
Measure: Count of Units; unit: eyelids
Units Other Than Participants: eyelids
Arm/Group | BRAP (Bevel/Rotate/Advance Procedure) | Trabut 3 mm
Number analyzed (Participants) | 335 | 328
Number analyzed (eyelids) | 425 | 420
eyelids | 3 | 10

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through 10-20-month follow-up.
Arm/Group | BRAP (Bevel/Rotate/Advance Procedure) | Trabut 3 mm
All-Cause Mortality (participants affected / at risk) | 7/351 | 6/349
Serious Adverse Events (participants affected / at risk) | 0/351 | 0/349
Other Adverse Events (participants affected / at risk) | 0/351 | 0/349

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT03886519/Prot_SAP_000.pdf